CLINICAL TRIAL: NCT01390961
Title: Comparison of Tolerability Between Two Allergy Drops
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hom, Milton M., OD, FAAO (Individual)
Collaborators: Allergan (Industry)
Responsible Party: Milton M. Hom, OD, FAAO., Private Practice
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IIT-000256
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-07

CONDITIONS: Allergic Conjunctivitis
Keywords: Allergic conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Naphazoline; Pheniramine; alcaftadine; Naphcon A

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: alacaftadine and naphazoline HCl & pheniramine maleate — once a day
  Other Names: Lastacaft; Opcon A

SUMMARY:
Comfort is compared between two allergy drops

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and over inclusive.
* Males or females
* Patient is in generally good & stable overall health.
* Patient likely to comply with study guidelines & study visits.
* Informed consent signed.
* History of allergic conjunctivitis
* Current symptoms of allergic conjunctivitis assessed by the investigator

Exclusion Criteria:

* Corneal refractive surgery or contact lens wear within 6 months of this study.
* Current use of Restasis
* Intra-ocular surgery within 6 months or ocular laser surgery within 6 months.
* Pregnant or lactating women.
* Ocular pathology (includes glaucoma and cataract), which could impact results and/or place patient at risk.

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-12 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Tolerability | 8 weeks
  Tolerability measured by questionnaire Visual Analog scale 1 to 100

CONTACTS AND LOCATIONS:
Locations (1):
- Milton M. Hom, OD, FAAO., Azusa, California, United States